CLINICAL TRIAL: NCT00304876
Title: Fecal Bacterial Flora in Clostridium Difficile-Associated Diarrhea
Status: Completed | Type: Observational
Sponsor: Michael E. DeBakey VA Medical Center (U.S. Federal Agency)
Collaborators: Baylor College of Medicine (Other)
Responsible Party: Daniel Musher, MD, VAHouston
Other Study IDs: H-18158
Record Dates: First submitted 2006-03-16; First posted 2006-03-20 (Estimated); Last update posted 2010-09-10 (Estimated); Status verified 2010-09

CONDITIONS: Enterocolitis; Pseudomembranous Colitis; Antibiotic-Associated Colitis
Keywords: Clostridium difficile associated diarrhea
MeSH Terms: conditions — Enterocolitis; Enterocolitis, Pseudomembranous

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The investigators propose to study intensively the bacteriology of feces in C. difficile associated diarrheal disease, using a variety of conventional and very up-to-date techniques.

DETAILED DESCRIPTION:
Clostridium difficile associated colitis is an increasing problem in hospitals throughout the developed world; the number of cases has increased, and the failure to respond to conventional therapy has become far more common. The investigators have recently documented in the medical literature (Clin Infect Dis, June, 2005; Lancet Infect Dis, August, 2005). Possible reasons for failure of treatment include persistence of C. difficile and/or imbalance of other bacterial flora in the colon. The bacteriology of fecal flora in C. difficile associated diarrhea has not been studied.

ELIGIBILITY:
Inclusion Criteria:

* Patients with antibiotic-associated diarrhea with a positive assay for C. difficile toxin
* Patients with antibiotic-associated diarrhea with 3 negative assays for C. difficile toxin
* Patients with antibiotic-associated diarrhea that has failed to respond to conventional therapy
* Hospitalized patients who have received >2 antibiotics and who have no symptoms of diarrhea or abdominal discomfort

Exclusion Criteria:

* none

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients positive for C. difficile
Sampling Method: Non-Probability Sample
Enrollment: 5 (Actual)
Dates: Start 2005-10; Primary Completion 2007-01 (Actual); Study Completion 2007-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Daniel M Musher, M.D., Principal Investigator — Baylor College of Medicine, Houston VA Medical Center
Locations (2):
- United States (2):
  - Johns Hopkins Medical Research Institute, Baltimore, Maryland
  - Michael E. DeBakey Veterans Affairs Medical Center, Houston, Texas